CLINICAL TRIAL: NCT05248893
Title: A Phase 3, Multicenter, Open-label Study to Evaluate the Safety of AGN-151586 for the Treatment of Glabellar Lines
Brief Title: A Study to Assess Adverse Events of Intramuscular AGN-151586 Injection in Adult Participants With Glabellar Lines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M21-509
Record Dates: First submitted 2022-02-14; First posted 2022-02-21 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Glabellar Lines
Keywords: Glabellar Lines; AGN-151586

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- AGN-151586 (Experimental): Participants will receive 5 intramuscular injections in the glabellar complex on Day 1. Based on meeting the retreatment criteria, the participant may receive up to 2 additional cycles of open-label treatments.
  Interventions: Drug: AGN-151586

INTERVENTIONS:
Drug: AGN-151586 — Intramuscular Injection

SUMMARY:
Facial lines that develop from repeated facial expression, such as glabellar lines (GL), are typically treated by selectively weakening specific muscles with small quantities of botulinum toxin. The purpose of this study is to evaluate the safety of AGN-151586 over multiple repeat treatments of the study drug to improve the appearance of glabellar lines.

AGN-151586 is an investigational product being developed for the treatment of GL. Around 940 to 1100 adult participants with moderate to severe GL will be enrolled in the study in approximately 45 sites in the United States.

This is an open-label, 126 day study in which all participants will receive 5 intramuscular AGN-151586 injections to the glabellar complex on Day 1. Participants meeting retreatment criteria may receive up to 2 additional cycles of treatment during the study.

Participants will attend regular visits during the study at a study site. The effect of the treatment will be checked by medical assessments, blood tests, telephone calls, questionnaires and checking for side effects.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be able to accurately assess their facial lines without the use of eyeglasses (contact lens use is acceptable).
* Participant must have moderate or severe Glabellar Lines at maximum frown as assessed by both the investigator and participant using the Facial Wrinkle Scale (FWS) at Screening and Baseline Day 1 visit.

Exclusion Criteria:

* Uncontrolled systemic disease.
* Presence or history of any medical condition that may place the subject at increased risk following exposure to AGN-151586 or interfere with the study evaluation, including:

  * Diagnosed myasthenia gravis, Lambert-Eaton syndrome, amyotrophic lateral sclerosis, or any other significant disease that might interfere with neuromuscular function
  * History of facial nerve palsy
  * Infection or dermatological condition at the treatment injection sites
  * Marked facial asymmetry, dermatochalasis, deep dermal scarring, excessively thick sebaceous skin, excessively photodamaged skin, or the inability to substantially lessen facial lines even by physically spreading them apart
  * Any eyebrow or eyelid ptosis at screening or Baseline Day 1 visit as determined by the investigator
* History of known immunization to any botulinum toxin serotype.
* Participants who have reported use of any botulinum neurotoxin of any serotype (including any investigational botulinum neurotoxin product) for aesthetic treatment within the last 6 months prior to screening and for therapeutic treatment within the last 12 months prior to study drug administration.
* Tattoos, jewelry, or clothing which obscure the glabellar area and cannot be removed.
* Anticipated need for surgery or overnight hospitalization during the study.
* History of surgical procedures on forehead and/or periorbital areas or affecting these areas including any lifting procedure (e.g., rhinoplasty, facial lift, suture lift, thread lift, brow lift, eyelid and/or eyebrow surgery).
* History of periorbital, mid-facial, or upper-facial treatment with semi-permanent or permanent soft tissue fillers (e.g., poly-L-lactic acid, polyalkylimide, polymethylmethacrylate, polytetrafluoroethylene, and silicone), synthetic implantation and/or autologous fat transplantation.
* Known active severe acute respiratory syndrome coronavirus 2 (SARSCoV-2) infection.
* Female subject who is pregnant or breastfeeding, and is considering becoming pregnant or donating eggs during the study or for approximately 30 days after the last dose of study drug or until the end of study, whichever is longer.
* Participant who has been treated with any investigational drug within 30 days or 5 half-lives of the drug (whichever is longer) prior to the first dose of study drug or is currently enrolled in another clinical study or was previously enrolled in this study.
* Anticipated need for treatment with botulinum neurotoxin of any serotype for any reason during the study (other than study drug).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 986 (Actual)
Dates: Start 2022-02-25 (Actual); Primary Completion 2023-06-26 (Actual); Study Completion 2023-06-26 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | Day 1 to Day 126
  An adverse event (AE) is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with the treatment. The investigator assesses the relationship of each event to the use of study drug.
Change in Vital Sign Measurements | Day 1 to Day 126
  Percentage of participants with abnormal change from baseline in vital sign measurements like systolic and diastolic blood pressure will be assessed.
Change in Electrocardiogram (ECG) Measurements | Day 1 to Day 126
  12-lead resting ECGs will be recorded. Parameters include heart rate, PR interval, QT interval, QRS duration, and QT interval corrected using Fridericia's formula (QTcF).
Presence of binding and neutralizing antidrug antibodies | Day 1 to Day 126
  Blood samples for immunogenicity testing will be collected from all participants treated with AGN-151586 at predetermined timepoints. Collected samples will be processed to yield serum for detection of binding and neutralizing antibodies to AGN-151586.

CONTACTS AND LOCATIONS:
Overall Officials: ALLERGAN INC., Study Director — Allergan
Locations (43):
- United States (41):
  - Skin Wellness Dermatology - Homewood /ID# 241233, Birmingham, Alabama
  - Advanced Research Associates - Glendale /ID# 232245, Glendale, Arizona
  - Skin Care and Laser Physicians of Beverly Hills /ID# 241237, Los Angeles, California
  - The Eye Research Foundation /ID# 232229, Newport Beach, California
  - Cosmetic Laser Dermatology /ID# 243513, San Diego, California
  - UC San Diego Health - University Center Lane - La Jolla /ID# 241243, San Diego, California
  - Ava T. Shamban MD - Santa Monica. /ID# 241246, Santa Monica, California
  - Art of Skin MD /ID# 241244, Solana Beach, California
  - Moradi MD /ID# 241242, Vista, California
  - AboutSkin Research, LLC /ID# 241702, Greenwood Village, Colorado
  - Susan H. Weinkle MD /ID# 233835, Bradenton, Florida
  - Skin Research Institute LLC /ID# 232240, Coral Gables, Florida
  - Skin and Cancer Associates, LLP /ID# 232228, Miami, Florida
  - ForCare Clinical Research /ID# 241229, Tampa, Florida
  - Hamilton Research, LLC /ID# 241232, Alpharetta, Georgia
  - Atlanta Biomedical Clinical Research /ID# 241258, Atlanta, Georgia
  - Meridian Clinical Research Dermatology /ID# 241234, Savannah, Georgia
  - DeNova Research /ID# 232231, Chicago, Illinois
  - Advanced Dermatology /ID# 241252, Lincolnshire, Illinois
  - Laser and Skin Surgery Center of Indiana /ID# 233834, Indianapolis, Indiana
  - Coleman Center For Cosmetic Dermatologic Surgery /ID# 232230, Metairie, Louisiana
  - Etre Cosmetic Dermatology and Laser Center /ID# 232235, New Orleans, Louisiana
  - Visage Dermatology and Aesthetic Center /ID# 241248, Largo, Maryland
  - Rkmd, Llc /Id# 241239, North Bethesda, Maryland
  - Michigan Center for Research Company /ID# 241255, Clarkston, Michigan
  - Rao Dermatology /ID# 243515, Atlantic Highlands, New Jersey
  - image Dermatology, P.C. /ID# 241227, Montclair, New Jersey
  - The Rejuva Center /ID# 244285, Latham, New York
  - Mariwalla Dermatology /ID# 241240, West Islip, New York
  - Northwest Dermatology Institute /ID# 233498, Portland, Oregon
  - Perelman Center for Advanced Medicine - /ID# 243966, Philadelphia, Pennsylvania
  - Sherman Aesthetic Center /ID# 241247, Nashville, Tennessee
  - Tennessee Clinical Research Center /ID# 241254, Nashville, Tennessee
  - DermResearch, Inc. Austin, TX /ID# 241228, Austin, Texas
  - Bellaire Dermatology Associates /ID# 232243, Bellaire, Texas
  - J&S Studies, Inc. /ID# 241236, College Station, Texas
  - Dallas Center for Dermatology and Aesthetics /ID# 241245, Dallas, Texas
  - Swinyer-Woseth Dermatology /ID# 241250, Salt Lake City, Utah
  - The Education & Research Foundation, Inc. /ID# 241225, Lynchburg, Virginia
  - Premier Clinical Research /ID# 233836, Spokane, Washington
  - EthiQ2 Research, LLC /ID# 241256, Brookfield, Wisconsin
- Puerto Rico (2):
  - Santa Cruz Behavioral (SCB) Research Center /ID# 241226, Bayamón
  - Jose Raul Montes Eyes & Facial Rejuvenation-Torre Medica Aux /ID# 241241, San Juan

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/